CLINICAL TRIAL: NCT03234491
Title: Improving Post-Prandial Blood Glucose Control With Afrezza During Closed-Loop Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2000020715
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Post-Prandial Hyperglycemia; Post-Prandial Hypoglycemia
Keywords: Diabetes; Insulin
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- A-HCL low (Active Comparator): Trial arms will entail (a) HCL with RAI analog (insulin lispro or aspart) pre-meal bolus (R-HCL visit), (b) ACL with pre-meal dose titrated down to the lower dose inhaled insulin (AHCL low visit), and (c) ACL with pre-meal dose titrated up to higher dose inhaled insulin (A-HCL high visit).
  Interventions: Device: DiAS; Drug: Afrezza low dose
- A-HCL high (Active Comparator): Trial arms will entail (a) HCL with RAI analog (insulin lispro or aspart) pre-meal bolus (R-HCL visit), (b) ACL with pre-meal dose titrated down to the lower dose inhaled insulin (AHCL low visit), and (c) ACL with pre-meal dose titrated up to higher dose inhaled insulin (A-HCL high visit).
  Interventions: Device: DiAS; Drug: Afrezza high dose
- R-HCL (Active Comparator): Trial arms will entail (a) HCL with RAI analog (insulin lispro or aspart) pre-meal bolus (R-HCL visit), (b) ACL with pre-meal dose titrated down to the lower dose inhaled insulin (AHCL low visit), and (c) ACL with pre-meal dose titrated up to higher dose inhaled insulin (A-HCL high visit).
  Interventions: Device: DiAS

INTERVENTIONS:
Device: DiAS — Diabetes Assistant (DiAS) hybrid closed loop system.
Drug: Afrezza low dose — Afrezza inhaled insulin low dose.
  Arms: A-HCL low
Drug: Afrezza high dose — Afrezza inhaled insulin high dose.
  Arms: A-HCL high

SUMMARY:
The study will be conducted in two phases; an in-patient meal study phase (Phase I) and an outpatient home study (Phase II). The two phase study design is chosen to enhance safety by testing the Afrezza Closed-Loop (CL) system in controlled in-clinic setting under study staff supervision before it could be investigated at the outpatient home setting. Phase II will not begin without the establishment of safety in Phase I.

DETAILED DESCRIPTION:
There are 2 primary study aims that this research will address. The first study aim will be to determine whether use of Afrezza inhaled insulin with ultra-fast kinetics will improve the performance of a closed-loop (CL) system, both with respect to immediate post-prandial hyperglycemia and the subsequent late post-prandial hypoglycemia as compared to hybrid CL (HCL) with subcutaneous (SC) rapid-acting insulin (RAI) pre-meal bolus.

The second study aim will be to examine the efficiency and feasibility of Afrezza inhaled insulin as a pre-meal bolus and a missed meal correction bolus on mitigating post-prandial blood glucose control during outpatient CL therapy.

This study will test the hypothesis that Afrezza inhaled insulin given before a meal to mimic physiologic first phase insulin release will limit the magnitude and rate of rise of glucose levels following a meal and will achieve greater percent time spent within target blood glucose range as compared to conventional hybrid CL therapy without inhaled insulin both in the in-clinic research and outpatient real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* The age inclusion criterion is 18-29 years for phase I and 18-50y for phase II
* Previously diagnosed with Type 1 Diabetes Mellitus, as determined by the judgment of the Principal Investigator, based on clinical presentation and as documented in the clinic record (formal antibody or genetic testing will not be required).
* Diabetes duration at least 1 year.
* Willing to have an intravenous (IV) line inserted for frequent blood sampling and infusion of glucose.
* Hemoglobin A1c (HbA1c) ≤10%
* Speak and understand English.

Exclusion Criteria:

* HbA1c >10.0% at the time of screening
* Insulin pump naïve subjects and subjects with unstable insulin dosing parameters requiring daily adjustments in insulin sensitivity factor, insulin to carbohydrate ratio and basal rates other than the established temporary rates that are determined to manage specific conditions such as exercise.
* History of an episode of severe hypoglycemia or Diabetic Ketoacidosis (DKA) requiring inpatient management within six months prior to the screening visit and/or subjects with history of clinician diagnosed hypoglycemia unawareness.
* History of recurrent DKA defined as more than three episodes of admissions for DKA during the past 12 months.
* Subjects requiring an insulin total daily dose <0.1u/kg/day and >3u/kg/day.
* History of physician diagnosis of asthma or any other clinically important pulmonary disease, or use of any medications to treat such conditions within the last year
* Allergy or know hypersensitivity for Afrezza or to drugs with similar chemical structure
* Any disease or exposure to any medication which, in the judgment of the principal investigator, may impact glucose metabolism.
* FEV1 <70% of NHANES III; Forced vital capacity (FVC) < 70% of NHANES III predicted for children ≥8 years of age.
* Positive urine pregnancy test for female patients of childbearing, breast feeding, or intention to become pregnant.
* Smoking of tobacco or other substances.
* Subjects who discontinued smoking (including cigarettes, cigars, pipes) within the past 6 months.
* History of abnormal spirometry or chest X-ray suggestive of lung disease.
* History of respiratory tract malignancy.
* Any condition or medication that may result in pulmonary toxicity (e.g. current or previous chemotherapy or radiation therapy or history of or current use of amiodarone).
* Inability to perform study procedures including pulmonary function testing and Afrezza inhalation using the BluHale system.
* Patients who take acetaminophen containing medications on a regular basis or anticipate taking during the study period and are unable and/or unwilling to substitute with a non-acetaminophen containing medication.
* Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the DexCom CGM (implantable cardioverter defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants).
* Active gastroparesis requiring current medical therapy.
* Known bleeding diathesis or dyscrasia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
PostPrandial Blood Glucose | Up to 4 hours following meal
  Continuous glucose monitoring (CGM) using Yellow Springs Instrument (YSI) will be used to measure blood glucose (mg/dl). Data will be collected for a maximum 4 hours following each meal.

SECONDARY OUTCOMES:
Insulin Levels | Up to 4 hours following meal
  Insulin levels will be monitored during the study. It will will be calculated and reported by each one of the three treatment groups with the appropriate metric (mean(SD) or median(IRQ)).
Venous Glucose Levels | Up to 4 hours following meal
  The changes in venous levels from t=0 to peak and the peaks will be calculated and reported by each one of the three treatment groups with the appropriate metric (mean(SD) or median(IRQ)).

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Diabetes Research Clinic, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Galderisi A, Cohen N, Calhoun P, Kraemer K, Breton M, Weinzimer S, Cengiz E. Effect of Afrezza on Glucose Dynamics During HCL Treatment. Diabetes Care. 2020 Sep;43(9):2146-2152. doi: 10.2337/dc20-0091. Epub 2020 Jul 13. PMID 32661108